CLINICAL TRIAL: NCT03759912
Title: The Efficacy of Ultra-High-Resolution Mapping Guided Partial Antral Ablation for Atrial Fibrillation
Brief Title: Ultra-High-Resolution Mapping Guided Partial Antral Ablation for AF
Acronym: TAILOR
Status: Terminated | Type: Observational
Why Stopped: The trial stopped prematurely because of enrollment challenges.
Sponsor: Keimyung University Dongsan Medical Center (Other)
Collaborators: Boston Scientific Corporation (Industry)
Responsible Party: Principal Investigator, Seongwook Han, Professor, Keimyung University Dongsan Medical Center
Other Study IDs: 2018-07-008
Record Dates: First submitted 2018-11-25; First posted 2018-11-30 (Actual); Last update posted 2023-05-31 (Actual); Status verified 2023-05

CONDITIONS: Atrial Fibrillation
Keywords: Atrial fibrillation ablation; Pulmonary vein; Ultra high resolution mapping
MeSH Terms: conditions — Atrial Fibrillation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- PVI using Ultra-High-Resolution Mapping: The paroxysmal atrial fibrillation patients who received pulmonary vein antral catheter ablation for electrical isolation of pulmonary veins using ultra-high-resolution mapping system (Rhythmia High Density mapping system).

SUMMARY:
The electrical isolation of the pulmonary veins (PVI) is the cornerstone of current ablation techniques for the treatment of atrial fibrillation (AF) because the PV is the most common trigger of AF. Wide bi-antral circumferential ablation (WACA) is more effective than segmental PV isolation in achieving freedom from total atrial tachyarrhythmia recurrence at long-term follow-up. Therefore, it is widely accepted as initial ablation strategy. However, the WACA technique requires a much larger number of ablation and higher energy to achieve complete isolation because of thick atrial myocardial sleeves with multiple muscle layers present in most of the PV antrum, which is less likely to achieve homogenous transmural lesions in the entire circumference with the currently available ablation technologies. Meanwhile, muscular discontinuities and abrupt changes of the fiber orientation in human PV-Left atrium (LA) junction are previously reported, and electrical PV isolation can usually be achieved without complete circumferential ablation. However, the current electroanatomical mapping (EAM) system has a limitation to understand the complex relationship of PV-LA junction mainly due to relatively low resolution.

The Rhythmia mapping system (BostonScientific, Inc, Cambridge, MA) is a new system provides ultra-high-resolution EAM using a small basket array of 64 electrodes (IntellaMap Orion, Boston Scientific). Owing to better resolution, this new system capable of rapidly and accurately identify critical isthmuses and low-voltage regions of interest and also allows automatic acquisition and accurate annotation of the electrograms, without the need for manual correction.

In this context, we hypothesized that rapid and precise identification of activation pattern of PV-LA junction by Rhythmia system could allow complete, durable electrical isolation of PVs without circumferential antral ablation.

ELIGIBILITY:
Inclusion Criteria:

1. Age over 20 years old and under 80 years old
2. Patients with non-valvular paroxysmal atrial fibrillation
3. Patients having atrial fibrillation even after receiving continued treatment with at least 1 antiarrhythmic drug for more than 6 weeks
4. Patients who could have informed consent
5. Patients who are available for a follow-up of more than at least three months after the catheter ablation

Exclusion Criteria:

1. Patients unsuitable for catheter ablation due to a previous history of pulmonary surgery or structural heart disease
2. Patients who cannot receive standard treatments such as anticoagulation therapy needed before the radiofrequency catheter ablation
3. Patients in the subject group vulnerable to a clinical study
4. Patients who had undergone a prior catheter ablation for atrial fibrillation

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Paroxysmal atrial fibrillation patients who received pulmonary vein isolation using Rhythmia HDx mapping system in Keimyung University Dongsan Medical Center.
Sampling Method: Non-Probability Sample
Enrollment: 75 (Actual)
Dates: Start 2018-11-20 (Actual); Primary Completion 2020-08-05 (Actual); Study Completion 2021-08-07 (Actual)

PRIMARY OUTCOMES:
Atrial arrhythmia recurrence | one year
  recurrence of atrial tachyarrhythmia after the index procedure

SECONDARY OUTCOMES:
acute pulmonary vein isolation rate | During procedure
  Percentage of patients who are able to obtain pulmonary vein isolation during the procedure
acute pulmonary vein reconnection rate | During procedure
  Percentage of patients who achieve pulmonary vein isolation during the procedure but have PV reconnection within the procedure
percentage of ablation area in the antrum | During procedure
  Area of pulmonary vein antrum ablated to obtain pulmonary vein isolation
Procedural outcome | During procedure
  procedure time in minute
Procedural outcome | During procedure
  fluoroscopic time in minute
Procedural outcome | During procedure
  total ablation time in minute
Procedural outcome | During procedure
  procedural complications - number of patients who experienced complications

CONTACTS AND LOCATIONS:
Overall Officials: Seongwook Han, MD, PhD, Principal Investigator — Keimyung University
Locations (1):
- Keimyung University Dongsan Medical Center, Daegu, South Korea